CLINICAL TRIAL: NCT00600119
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Multiple-Dose, Dose Escalation Study to Evaluate the Efficacy, Safety and Tolerability of NKTR-118 in Patients With Opioid-Induced Constipation (OIC)
Brief Title: A Phase 2, Double-Blind, Multiple-Dose Escalation Study to Evaluate NKTR-118 (Oral PEG-Naloxol) in Patients With Opioid-Induced Constipation (OIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-IN-NX003
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Opioid Induced Constipation (OIC)
Keywords: NKTR, constipation, opioid, induced, bowel, dysfunction, Naloxol, Naloxone, Narcan, PEG naloxol, OIC, OBD, Nektar
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- B (Experimental): NKTR-118
  Interventions: Drug: NKTR-118

INTERVENTIONS:
Drug: placebo — placebo, oral, once daily (QD)
  Arms: A
Drug: NKTR-118 — 5 mg, 25 mg, 50 mg or 100 mg, oral,once daily (QD)
  Arms: B

SUMMARY:
Study (07-IN-NX003) is a Phase 2, multi-center, placebo-controlled, double-blind, randomized, dose-escalation trial. It is designed to investigate the safety, efficacy and tolerability of NKTR-118 (PEG-naloxol) in patients with opioid-induced constipation (OIC) and other clinical manifestations of opioid-induced bowel dysfunction (OBD). The objective of this study is to evaluate the safety, effectiveness and pharmacokinetics of NKTR-118 at 4 different doses.

ELIGIBILITY:
Main Inclusion Criteria:

* 18 years of age or older, male or female
* Receiving a stable opioid regimen
* Documented opioid-induced constipation
* Willingness to stop all laxatives and other bowel regimens. The use of constipation rescue medication will be allowed during the study.

Main Exclusion Criteria:

* Life expectancy less than 6 months
* Active substance abuse
* Fecal incontinence, irritable bowel syndrome, inflammatory bowel disease, or other active medical disorders associated with diarrhea or intermittent loose stools or constipation
* Pregnant or breast-feeding
* Any receipt of an investigational medication within 30 days of screening
* History or presence of specific cardiac, neurologic, endocrine and/or psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, Study Director — AstraZeneca Pharmaceuticals, Wilm DE
Locations (33):
- United States (33):
  - Tennessee Valley Pain Consultants / Center for Pain Management, Huntsville, Alabama
  - Deerfoot Internal Medicine, Pinson, Alabama
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Therapeutic Research Institute of Orange County, Laguna Hills, California
  - San Diego Managed Care Group, San Diego, California
  - Arapahoe Gastroenterology, PC, Littleton, Colorado
  - Southeast Clinical Research, Chiefland, Florida
  - Osler Medical, Inc. / Osler Clinical Research, Melbourne, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Gold Coast Research LLC, Weston, Florida
  - PMI Health Research Group, Atlanta, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Pain & Rehabilitation Clinic of Chicago, Chicago, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Gulf Coast Reserach, Baton Rouge, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - MAPS Applied Research Center, Edina, Minnesota
  - Midwest Pharmaceutical Research, Inc., City of Saint Peters, Missouri
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Four Seasons Hospice and Palliative Care, Flat Rock, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Riverhills Healthcare Research Division, Cincinnati, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Medford Medical Clinic, Medford, Oregon
  - Anderson Gastroenterology Associates, LLC, Anderson, South Carolina
  - Singleton Health Center, Orangeburg, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Spokane Internal Medicine, Spokane, Washington

REFERENCES:
- See also: 07-IN-NX003 CSR Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1143&filename=07-IN-NX003_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Canada, Germany, Romania, and the United States between 04 January 2008 and 23 March 2009.
Pre-assignment Details: The study duration was up to 11 weeks, consisting of an initial screening period lasting up to 10 days, a 14-day OIC confirmation period, during which the OIC diagnosis was confirmed, a 7-day single-blind placebo run-in period, a 29-day double-blind treatment period, and a follow-up visit 2 weeks after the last dose of study drug.
Groups:
- Placebo 5 mg: Placebo for NKTR-118 5 mg QD, oral treatment
- NKTR-118 5 mg: NKTR-118 5 mg QD, oral treatment
- Placebo 25 mg: Placebo for NKTR-118 25 mg QD, oral treatment
- NKTR-118 25 mg: NKTR-118 25 mg QD, oral treatment
- Placebo 50 mg: Placebo for NKTR-118 50 mg QD, oral treatment
- NKTR-118 50 mg: NKTR-118 50 mg QD, oral treatment
Period: Single-blind Placebo run-in Period
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Started | 36 | 35 | 29 | 31 | 39 | 37
Completed | 32 | 33 | 27 | 30 | 37 | 35
Not Completed | 4 | 2 | 2 | 1 | 2 | 2
Not completed — Other - Not specified | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Inclusion/Exclusion Criteria Not Met | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Started | 32 | 33 | 27 | 30 | 37 | 35
Completed | 27 | 28 | 27 | 28 | 31 | 21
Not Completed | 5 | 5 | 0 | 2 | 6 | 14
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Inclusion/Exclusion Criteria Not Met | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Moderate to Severe Opioid Withdrawal | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 2 | 10
Period: Follow-up Period
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Started | 27 | 28 | 27 | 28 | 31 | 21
Completed | 26 | 28 | 27 | 28 | 31 | 20
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are summarized based on the MITT analysis population, which consisted of all randomized patients who received at least 1 dose of double-blind study treatment, had a baseline value and Visit 6 evaluable data (where Visit 6 was the Week 1 visit during the double-blind study treatment period).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg | Total
Number analyzed (Participants) | 31 | 31 | 27 | 29 | 37 | 30 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (12.0) | 50.3 (13.1) | 51.0 (13.2) | 51.8 (11.4) | 48.4 (10.2) | 49.6 (11.0) | 49.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 18 | 15 | 23 | 21 | 115
  Male | 12 | 12 | 9 | 14 | 14 | 9 | 70
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 27 | 28 | 23 | 26 | 31 | 25 | 160
  Black | 4 | 3 | 3 | 2 | 4 | 5 | 21
  Not Allowed to Ask | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hispanic/Latino | 0 | 0 | 1 | 0 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Spontaneous Bowel Movements (SBMs) Per Week During Week 1
Description: Change from baseline in SBMs/week during Week 1 was defined as SBMs/week during the first week of double-blind study medication (between Visit 4 and Visit 6) minus baseline SBMs/week. Baseline was defined as the average SBMs/week during the 2-week OIC screening period. An SBM was defined as a BM without the use of laxatives in the previous 24 hours as recorded in the e-diary.
Time Frame: Days 1 through 7
Population: The MITT analysis population consisted of all randomized patients who received at least 1 dose of double-blind study treatment, had a baseline value and Visit 6 evaluable data (where Visit 6 was the Week 1 visit during the double-blind study treatment period).
Measure: Mean (Standard Deviation); unit: Number of SBMs/week
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Number analyzed (Participants) | 31 | 31 | 27 | 29 | 37 | 30
Number of SBMs/week | 1.8 (2.4) | 2.6 (3.6) | 1.9 (2.5) | 3.6 (2.3) | 1.9 (5.2) | 4.4 (3.8)
Statistical Analysis 1: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.7781, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0020, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in SBMs/Week Across the 28-day Double-blind Period
Description: Change from baseline in SBMs/week across the 28-day double-blind period was calculated as SBMs/week during 28-day double-blind study treatment period minus baseline SBMs/week. Baseline was defined as the average SBMs/week during the 2-week OIC screening period.
Time Frame: Days 1 through 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of SBMs/week
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Number analyzed (Participants) | 31 | 31 | 27 | 29 | 37 | 30
Number of SBMs/week | 1.7 (1.9) | 2.3 (2.9) | 1.7 (2.2) | 3.2 (2.0) | 1.2 (2.0) | 4.6 (3.4)
Statistical Analysis 1: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.5118, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0022, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation-Quality of Life (PAC-QOL) Questionnaire
Description: The PAC-QOL scale is a 28-item self-report instrument designed to evaluate the burden of constipation on patients' everyday functioning and well-being in the 2 weeks (14 days) prior to assessment. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely).The instrument can be used to generate an overall score, but is also reported to assess 4 specific constipation-related domains including: 1) worries and concerns (11 items), 2) physical discomfort (4 items), 3) psychosocial discomfort (8 items), and 4) satisfaction (5 items). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items. The range is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). A negative change from baseline indicates improvement.
Time Frame: Days 1 through 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Number analyzed (Participants) | 28 | 30 | 25 | 28 | 35 | 29
units on a scale
  Physical Discomfort domain | 1.4 (1.0) | 1.2 (0.8) | 1.7 (0.9) | 1.2 (1.0) | 1.7 (1.1) | 1.3 (1.0)
  Worries/Concerms domain | 1.5 (1.1) | 1.3 (0.9) | 1.6 (1.1) | 1.1 (0.9) | 1.5 (1.0) | 1.2 (0.8)
  Psychosocial Discomfort domain | 0.8 (0.7) | 0.8 (0.8) | 1.1 (1.0) | 0.8 (0.8) | 1.0 (0.9) | 0.8 (0.8)
  Satisfaction domain | 2.6 (1.1) | 2.4 (1.1) | 2.8 (0.9) | 2.0 (1.3) | 2.8 (1.1) | 2.2 (1.1)
  Total Score | 1.5 (0.8) | 1.3 (0.8) | 1.7 (0.8) | 1.2 (0.8) | 1.6 (0.8) | 1.3 (0.8)
Statistical Analysis 1: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.5522, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Physical Discomfort domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 2: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0589, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Physical Discomfort domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 3: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.1691, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Physical Discomfort domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 4: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.6293, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Worries/Concerns domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 5: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0836, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Worries/Concerns domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 6: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.1155, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Worries/Concerns domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 7: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.9938, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Psychosocial Discomfort domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 8: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.2101, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Psychosocial Discomfort domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 9: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.4597, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Psychosocial Discomfort domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 10: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.4822, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Satisfaction domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 11: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0171, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Satisfaction domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 12: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.0160, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Satisfaction domain from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 13: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.6857, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Total Score from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 14: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0253, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Total Score from Baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 15: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.0772, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-QOL Total Score from Baseline (Week 1) to end of treatment (Week 4)

4. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation-Symptoms (PAC-SYM) Questionnaire
Description: The PAC-SYM questionnaire is a 12-item questionnaire that evaluates the severity of symptoms of constipation in 3 domains (stool, rectal, and abdominal symptoms) on a 5-point Likert scale ranging from 0 (absent) to 4 (very severe) in the 2 weeks (14 days) prior to assessment. Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items (ie, symptoms). The range is 0 (response is 'absent' for each item) to 4 (response is 'very severe' for each item). A negative change from baseline indicates improvement.
Time Frame: Days 1 through 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo 5 mg | NKTR-118 5 mg | Placebo 25 mg | NKTR-118 25 mg | Placebo 50 mg | NKTR-118 50 mg
Number analyzed (Participants) | 28 | 30 | 25 | 28 | 35 | 29
units on a scale
  Abdominal Symptoms domain | 1.2 (0.8) | 1.1 (0.9) | 1.4 (0.9) | 1.1 (0.9) | 1.2 (1.0) | 1.3 (1.0)
  Rectal Symptoms domain | 0.7 (0.8) | 0.7 (0.7) | 0.8 (0.8) | 0.7 (0.8) | 1.2 (1.0) | 0.7 (0.8)
  Stool Symptoms domain | 1.5 (1.0) | 1.5 (0.8) | 1.7 (0.8) | 1.2 (0.9) | 1.8 (1.1) | 1.2 (0.9)
  Total Score | 1.2 (0.8) | 1.2 (0.7) | 1.4 (0.6) | 1.1 (0.8) | 1.5 (1.0) | 1.1 (0.9)
Statistical Analysis 1: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.5008, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Abdominal Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 2: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.1823, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Abdominal Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 3: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.7045, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Abdominal Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 4: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.7088, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Rectal Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 5: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.5828, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Rectal Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 6: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.0116, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Rectal Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 7: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.7848, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Stool Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 8: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0335, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Stool Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 9: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.0591, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Stool Symptoms domain from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 10: Comparison: Placebo 5 mg vs NKTR-118 5 mg; Test type: Superiority or Other; p = 0.9317, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Total Score from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 11: Comparison: Placebo 25 mg vs NKTR-118 25 mg; Test type: Superiority or Other; p = 0.0675, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Total Score from baseline (Week 1) to end of treatment (Week 4)
Statistical Analysis 12: Comparison: Placebo 50 mg vs NKTR-118 50 mg; Test type: Superiority or Other; p = 0.1745, Wilcoxon (Mann-Whitney) — Analysis for change in PAC-SYM Total Score from baseline (Week 1) to end of treatment (Week 4)

ADVERSE EVENTS:
Arm/Group | NKTR-118 25 mg | NKTR-118 5 mg | NKTR-118 50 mg | Placebo 25 mg | Placebo 5 mg | Placebo 50 mg
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/33 | 1/35 | 0/27 | 1/32 | 1/37
Other Adverse Events (participants affected / at risk) | 19/30 | 18/33 | 26/35 | 15/27 | 15/32 | 13/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 25 mg (N=30) | NKTR-118 5 mg (N=33) | NKTR-118 50 mg (N=35) | Placebo 25 mg (N=27) | Placebo 5 mg (N=32) | Placebo 50 mg (N=37)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 25 mg (N=30) | NKTR-118 5 mg (N=33) | NKTR-118 50 mg (N=35) | Placebo 25 mg (N=27) | Placebo 5 mg (N=32) | Placebo 50 mg (N=37)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (12) | 1 (1) | 6 (9) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (4) | 6 (6) | 9 (10) | 1 (1) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 5 (5) | 11 (11) | 1 (1) | 5 (5) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 3 (5) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 5 (7) | 7 (7) | 5 (5) | 2 (2) | 3 (3)
VOMITING (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 2 (2)
CHILLS (General disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
PAIN (General disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 4 (5) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 3 (3) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days